CLINICAL TRIAL: NCT05771142
Title: Evaluation of an Innovative Smart T-shirt Capable to Monitor ECG Signal and Related Parameters Through the Comparison With a Holter ECG and a Smartwatch
Acronym: Youcare
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bologna (Other)
Collaborators: AccYouRate S.p.A. (Unknown)
Responsible Party: Principal Investigator, Claudio Borghi, Professor/Dean, University of Bologna
Other Study IDs: Smart_t-shirt_2021; 156/2022/Disp/AOUBo (Other: Comitato Etico di Area Vasta Emilia Centro della Regione Emilia-Romagna (CE-AVEC))
Record Dates: First submitted 2023-02-10; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-02

CONDITIONS: Cardiac Arrhythmias
Keywords: smart t-shirt; wearable; electrocardiogram
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Smart t-shirt, ECG Holter and smartwatch patients: 24h ECG Monitoring - All participants will wear the smart t-shirt, the ECG Holter and the smartwatch at the same time
  Interventions: Device: Smart t-shirt; Device: ECG Holter; Device: Smartwatch

INTERVENTIONS:
Device: Smart t-shirt — 24h ECG Monitoring with the smart t-shirt under study
Device: ECG Holter — 24h ECG Monitoring with ECG Holter
Device: Smartwatch — 24h ECG Monitoring with a smartwatch

SUMMARY:
Evaluation of an innovative smart t-shirt capable to monitor ECG signal and related parameters through the comparison with a Holter ECG and a smartwatch

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the biosignal (ECG) acquisition features of the smart t-shirt, developed by University of Bologna in collaboration with AccYouRate S.p.A., comparing it with a standard Holter ECG. Secondly, the study wants to compare the parameters related to ECG signal calculated by the smart t-shirt with those calculated by commercial smartwatches.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects agree to participate in the study and having dated and signed the informed consent form,
2. Subjects who have the capability to communicate, to make themselves understood, and to comply with the study's requirements,
3. Male or female aged ≥ 18 years and ≤ 90 years old,
4. Subjects with Cardiac electrophysiological (heart rhythm) pathologies or under screening for the assessment of possible cardiac electrophysiological pathologies.

Exclusion Criteria:

1. Subjects that for different reasons have difficulties to wear the sensorized t-shirt or the alternative sensorized chest band: Movement's impairments; Dermatological reaction to t-shirt fabric or materials,
2. Any medical or surgical condition that would limit the patient adhesion to the study protocol,
3. Severe obesity and sever underweight,
4. Subject that are not able to understand the scope of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in subjects with heart rhythm pathologies or under assessment of possible heart rhythm pathologies.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-03-27 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Electrocardiogram (ECG): Heart rate (beats per minute) | 24 hours
  Smart t-shirt and ECG Holter comparison
Electrocardiogram (ECG): RR interval (seconds) | 24 hours
  Smart t-shirt and ECG Holter comparison
Electrocardiogram (ECG): Qualitative distinction of P-waves, QRS-complexes, T-waves, and noise levels | 24 hours
  Smart t-shirt and ECG Holter comparison

SECONDARY OUTCOMES:
Electrocardiogram (ECG): Heart rate (beats per minute) | 24 hours
  Smart t-shirt and smartwatch comparison

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Sant'Orsola Malpighi - University of Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided